CLINICAL TRIAL: NCT01835613
Title: Evaluation Effects of Treatment With IL-6R Inhibitor on Clinical Response and Biomarkers in Patients With Rheumatoid Arthritis (RA) Not Responding to DMARDs and/or a First Biological Agent.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Osservatorio Epidemiologico GISEA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AR/BIOM
Record Dates: First submitted 2013-04-01; First posted 2013-04-19 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Rheumatoid Arthritis; Early RA; RA; IL-6; IL-6R; Inhibitor; Inhibition; Tocilizumab; Biomarkers; DMARDs; Biological; DAS; SDAI; AR/BIOM; OEG
MeSH Terms: conditions — Arthritis, Rheumatoid; Inhibition, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tocilizumab (Other): Biomarkers Measures
  At the routine visits (0, 3, 6, 12 and 18 months), a clinical evaluation will be made and samples collected for assaying the biomarkers.
  Interventions: Other: Biomarkers Measures

INTERVENTIONS:
Other: Biomarkers Measures — At the routine visits (0, 3, 6, 12 and 18 months), a clinical evaluation will be made and samples collected for assaying the biomarkers.

SUMMARY:
The purpose of this study is to assess the clinical response to IL-6 inhibition defined as Low Disease Activity (DAS44) <2.4) at the follow-up visit at 12 months and the correlation between the biomarkers and treatment response.

ELIGIBILITY:
Inclusion criteria:

* Signed informed consent form;
* Patients aged 18 - 75 years;
* RA classified in compliance with the 2010 ACR/EULAR criteria;
* Patients that have to suspend a previous treatment with DMARDs for total ineffectiveness or intolerance to drugs and/or patients that have not responded adequately to first-line combination DMARDs / biological treatment;
* Patients for which is indicated to start a treatment with an inhibitor of IL-6R for high values indicative of systemic inflammation (ESR>=28 mm/hour, PCR>5 mg/l , Fibrinogen >400 mg/dl and or Albumin <3.5 g/dl) and high disease activity (DAS>2.4), or contraindications to DMARDs use which make it necessary to take biological drug in monotherapy.
* Corticosteroids therapy stable (< = 7.5 mg)for at least four weeks;
* Joint symptoms for at least three but no more than 24 months from the screening visit;
* DAS44 >2.4 and/or SDAI >11
* Willing and able to comply with study procedures and timing.

Exclusion criteria:

* On going pregnancy or lactation;
* Severe active infections;
* Patients with other clinically significant concomitant diseases whose treatment or outcome could interfere with the expected evaluations of the study protocol.
* Blood AST or ALT levels >5 times the upper normal limit;
* ANC count <0.5 x 109/L
* Platelet count <50 x103 /μL
* Patients with other autoimmune rheumatic diseases, in addition to AR (for example systemic lupus erythematosus [SLE], scleroderma, polymyositis, ecc…)
* Medical history or concomitant joint diseases in additions to AR (for example tophaceous gout, reactive arthritis, psoriatic arthritis).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-07 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Disease Activity Score (DAS-44) | 12 months

SECONDARY OUTCOMES:
Simplified Disease Activity Index (SDAI);Biomarkers Measures | SDAI at 3-6-12-18 months
Biomarkers Measures | Biomarkers Measures at 3-6-12-18 months
  Evaluation by ELISA of the levels of the following biomarkers:
  IL-8, MCP-1, Chemerin, IL-1α, IL-1β, IL-17, IL-23, TGFβ1, IL-10, BAFF.in the plasma:

CONTACTS AND LOCATIONS:
Overall Officials: Gianfranco Ferraccioli, Prof., Principal Investigator — Dipartimento di Reumatologia, Università Cattolica del Sacro Cuore, Roma
Locations (1):
- Università Cattolica del Sacro Cuore, Roma, Italy